CLINICAL TRIAL: NCT00629070
Title: In Vivo Assessment of Quadriceps Muscle Plasticity in Children With Cerebral Palsy
Brief Title: Quadriceps Muscle Plasticity in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDS 087657
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; muscle strength; muscle architecture; ultrasound; rehabilitation; rectus femoris; quadriceps muscle
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ST (Experimental): Traditional strength training
  Interventions: Other: Traditional strength training
- VT (Experimental): Velocity-enhanced training
  Interventions: Other: Velocity-enhanced training

INTERVENTIONS:
Other: Traditional strength training — Performed 3 x week for 8 weeks on an isokinetic dynamometer (knee extension exercise)at 30 degrees/second; 6 sets of 5 maximum-effort concentric actions
  Arms: ST
Other: Velocity-enhanced training — Performed 3 x week for 8 weeks on an isokinetic dynamometer (knee extension exercise). Subjects will perform 2 sets of 5 concentric exertions at 30°/second. The following 4 sets of 5 repetitions will be performed at a faster speed, starting at 60° /second. The velocity will be increased weekly in 15° /second increments up to a maximum of 120°/second.
  Arms: VT

SUMMARY:
Our primary aim is to determine whether and how muscle architecture of the quadriceps muscles in cerebral palsy (CP) adapts to two separate training programs: traditional strength training (ST) vs. velocity-enhanced training (VT). For the ST group, we hypothesize that muscle size will increase in conjunction with strength. For the VT group, in addition to the above, we hypothesize that fiber length will increase with measures of muscle power. We also hypothesize that walking velocity will improve in both groups but that knee motion and step length will improve only with VT.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disability originating in childhood, occurring in 2-3 per 1,000 live births. Although the primary deficit in CP is injury to the brain, secondary impairments affecting muscle function such as weakness, contractures, and spasticity are often far more debilitating and lead to worsening disability throughout the lifespan. Some have suggested that these muscle changes in CP may be irreversible; however, it is now known that muscles are one of the most 'plastic' tissues in the body. In fact, recent evidence suggests that gross muscle hypertrophy and architectural changes within muscle fibers can occur as early as 3-5 weeks after resistance training in healthy adults. It is also unknown how effectively muscles in CP can adapt to training stimuli that target specific muscle architectural parameters, such as fascicle length and cross-sectional area. These parameters have been observed to be decreased in CP, suggesting loss of sarcomeres in-series (fiber shortening) and in-parallel (muscle atrophy). We propose here that specific training-induced muscle architectural adaptations can occur in CP, leading to improved motor function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Gross motor function classification system levels I, II, or III
* Ages 7 to 17

Exclusion Criteria:

* Orthopedic or neurosurgery within the past year
* Botulinum toxin injections within the 4 months prior to the study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-13 (Actual)

PRIMARY OUTCOMES:
Muscle thickness | before and after intervention

SECONDARY OUTCOMES:
Fascicle length | before and after intervention
Muscle strength (peak torque) | before and after intervention
Muscle power | before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Noelle G Moreau, PhD, PT, Principal Investigator — Medical University of South Carolina
Locations (1):
- Neuromuscular Assessment Laboratory, Charleston, South Carolina, United States

REFERENCES:
- [Background] Mohagheghi AA, Khan T, Meadows TH, Giannikas K, Baltzopoulos V, Maganaris CN. Differences in gastrocnemius muscle architecture between the paretic and non-paretic legs in children with hemiplegic cerebral palsy. Clin Biomech (Bristol). 2007 Jul;22(6):718-24. doi: 10.1016/j.clinbiomech.2007.03.004. Epub 2007 May 1. PMID 17475377
- [Background] Shortland AP, Harris CA, Gough M, Robinson RO. Architecture of the medial gastrocnemius in children with spastic diplegia. Dev Med Child Neurol. 2002 Mar;44(3):158-63. doi: 10.1017/s0012162201001864. PMID 12005316
- [Background] Damiano DL, Vaughan CL, Abel MF. Muscle response to heavy resistance exercise in children with spastic cerebral palsy. Dev Med Child Neurol. 1995 Aug;37(8):731-9. doi: 10.1111/j.1469-8749.1995.tb15019.x. PMID 7672470
- [Background] Moreau NG, Li L, Geaghan JP, Damiano DL. Contributors to fatigue resistance of the hamstrings and quadriceps in cerebral palsy. Clin Biomech (Bristol). 2009 May;24(4):355-60. doi: 10.1016/j.clinbiomech.2009.01.012. Epub 2009 Mar 5. PMID 19264384
- [Background] Moreau NG, Teefey SA, Damiano DL. In vivo muscle architecture and size of the rectus femoris and vastus lateralis in children and adolescents with cerebral palsy. Dev Med Child Neurol. 2009 Oct;51(10):800-6. doi: 10.1111/j.1469-8749.2009.03307.x. Epub 2009 Apr 21. PMID 19459913
- See also: Moreau Faculty web page — http://academicdepartments.musc.edu/chp/faculty/moreau.htm